CLINICAL TRIAL: NCT06436833
Title: Comparison of Bowel Preparation Using 2 Liter Polyethylene Glycol Regimen Plus Elobixibat Versus 4-Liter Polyethylene Glycol Regimen: a Randomized Controlled Trial
Brief Title: Comparison of Bowel Preparation Using 2 Liter Polyethylene Glycol Regimen Plus Elobixibat Versus 4-Liter Polyethylene Glycol Regimen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 67017
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-05

CONDITIONS: Bowel Preparation Solution; Colonoscopy
MeSH Terms: interventions — elobixibat

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2-Liter polyethylene glycol plus elobixibat (Experimental): Take Elobixibat 10 mg, one day before colonoscopy at 8 a.m. Take Polyethylene glycol 1 Liter, one day before colonoscopy at 8 p.m. Take polyethylene glycol 1 Liter, at day of colonoscopy at 5 a.m.
  Interventions: Drug: 2-Liter polyethylene glycol plus elobixibat
- 4-Liter polyethylene glycol (Active Comparator): Take Polyethylene glycol 2 Liter, one day before colonoscopy at 8 p.m. Take polyethylene glycol 2 Liter, at day of colonoscopy at 5 a.m.
  Interventions: Drug: 4-Liter polyethylene glycol

INTERVENTIONS:
Drug: 2-Liter polyethylene glycol plus elobixibat — Take Elobixibat 10 mg, one day before colonoscopy at 8 a.m. Take Polyethylene glycol 1 Liter, one day before colonoscopy at 8 p.m. Take polyethylene glycol 1 Liter, at day of colonoscopy at 5 a.m.
  Arms: 2-Liter polyethylene glycol plus elobixibat
Drug: 4-Liter polyethylene glycol — Take Polyethylene glycol 2 Liter, one day before colonoscopy at 8 p.m. Take polyethylene glycol 2 Liter, at day of colonoscopy at 5 a.m.
  Arms: 4-Liter polyethylene glycol

SUMMARY:
Comparison of bowel preparation using 2 liter polyethylene glycol regimen plus elobixibat Versus 4-Liter polyethylene glycol regimen. This study based on hypothesis that show Boston bowel preparation scale which 2L PEG regimen plus Elobixibat have result no significant difference from 4L PEG regimen

DETAILED DESCRIPTION:
The trial study in participant who visit to Rajavithi hospital for indication of colonoscopy such as Colorectal cancer screening, Iron deficiency anemia, Chronic diarrhea, chronic constipation, abdominal pain, unintentional weight loss, History of stool occult blood test , abnormal finding from imaging

Randomized participant as above in to two group as bowel preparation regimen Group 1 the participant recieved Polyethylene glycol 2 liter split dose plus Elobixibat 10 milligram.

Group 2 the participant recieved Polyethylene 4 liter split dose

Result of the study show the difference of 2 regimen of bowel preparation which regimen better than another by measuring cleanliness of bowel preparation. The cleanliness of bowel preparation measured by Boston bowel preparation scale

ELIGIBILITY:
Inclusion Criteria:

* Adute aged 18-80 year old
* Indication for colonoscopy(one selected)

  1. Colorectal cancer screening
  2. Stool occult blood test positive
  3. History of colonic polyp
  4. abdominal pain
  5. Iron deficiency anemia
  6. Chronic diarrhea
  7. chronic constipation
  8. Unintentional weight loss
  9. Gastrointestinal bleeding
  10. Abnormal imagind study
* Participant acceptconsent information

Exclusion Criteria:

* Pregnancy or lactation
* Gastroparesis, gastric outlet obstuction
* Bowel obstruction
* Gastrointestinal tract surgery
* Inflammatory bowel disease
* ASA(American society of anesthesiologist physical status) status > or = 4
* Allergic to Elobixibat or PEG
* Chronic kidney disease stage 4-5(GFR <30 ml/min)
* Biliary tract obstruction
* Previous history of inadequate bowel preparation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison efficacy of bowel preparation before colonoscopy between 2 group | During colonoscopy procedure
  Bowel preaparation measure by Boston bowel preparation scale

SECONDARY OUTCOMES:
Overall procedural time of colonoscopy | During colonoscopy procedure
  Duration since start colonoscopy insertion until withdrawal endoscope
Cecal intubation rate | During colonoscopy procedure
  Perform successful endoscopy to cecum
Withdrawal time of colonoscopy | During colonoscopy procedure
  Duration since endoscopy withdrawal from cecum to anal canal
Adenoma detection rate | During colonoscopy procedure
  At least one adenoma presented in this colonoscopy
Patient satisfaction in their bowel preparation regimen | 1 day before colonoscopy
  Satisfaction score evaluate by Linkert scale
Adverse event in each group | During 24 hour after taking bowel preparation
  Nausea, vomiting, abdominal pain, bloating, sleep disturbance, chest pain, dizziness, dyspnea, leg edema

CONTACTS AND LOCATIONS:
Overall Officials: Apichet Sirinawasatien, M.D., Study Chair — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
No plan for IPD sharing

REFERENCES:
- [Background] Yamaguchi D, Hidaka H, Matsunaga T, Akutagawa T, Tanaka Y, Jubashi A, Takeuchi Y, Tsuruoka N, Sakata Y, Miyahara K, Tominaga N, Kawakubo H, Takamori A, Shimoda R, Noda T, Ogata S, Tsunada S, Esaki M. Efficacy of elobixibat as bowel preparation agent for colonoscopy: Prospective, randomized, multi-center study. Dig Endosc. 2022 Jan;34(1):171-179. doi: 10.1111/den.14010. Epub 2021 May 24. PMID 33971037
- [Background] Nakajima A, Seki M, Taniguchi S. Determining an optimal clinical dose of elobixibat, a novel inhibitor of the ileal bile acid transporter, in Japanese patients with chronic constipation: a phase II, multicenter, double-blind, placebo-controlled randomized clinical trial. J Gastroenterol. 2018 Apr;53(4):525-534. doi: 10.1007/s00535-017-1383-5. Epub 2017 Aug 24. PMID 28840422
- [Background] Mohamed R, Hilsden RJ, Dube C, Rostom A. Split-Dose Polyethylene Glycol Is Superior to Single Dose for Colonoscopy Preparation: Results of a Randomized Controlled Trial. Can J Gastroenterol Hepatol. 2016;2016:3181459. doi: 10.1155/2016/3181459. Epub 2016 Apr 13. PMID 27446836
- [Background] Calderwood AH, Jacobson BC. Comprehensive validation of the Boston Bowel Preparation Scale. Gastrointest Endosc. 2010 Oct;72(4):686-92. doi: 10.1016/j.gie.2010.06.068. PMID 20883845
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] Parente F, Vailati C, Bargiggia S, Manes G, Fontana P, Masci E, Arena M, Spinzi G, Baccarin A, Mazzoleni G, Testoni PA. 2-Litre polyethylene glycol-citrate-simethicone plus bisacodyl versus 4-litre polyethylene glycol as preparation for colonoscopy in chronic constipation. Dig Liver Dis. 2015 Oct;47(10):857-63. doi: 10.1016/j.dld.2015.06.008. Epub 2015 Jul 6. PMID 26232311
- [Background] Acosta A, Camilleri M. Elobixibat and its potential role in chronic idiopathic constipation. Therap Adv Gastroenterol. 2014 Jul;7(4):167-75. doi: 10.1177/1756283X14528269. PMID 25057297
- [Background] Nakajima A, Taniguchi S, Kurosu S, Gillberg PG, Mattsson JP, Camilleri M. Efficacy, long-term safety, and impact on quality of life of elobixibat in more severe constipation: Post hoc analyses of two phase 3 trials in Japan. Neurogastroenterol Motil. 2019 May;31(5):e13571. doi: 10.1111/nmo.13571. Epub 2019 Feb 21. PMID 30793431
- [Background] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020